CLINICAL TRIAL: NCT00642811
Title: A Randomised, Double-Blind, Outpatient, Crossover Study of the Anti-platelet Effects of Ticagrelor Compared With Clopidogrel in Patients With Stable Coronary Artery Disease Previously Identified as Clopidogrel Non-responders or Responders [RESPOND]
Brief Title: A Study of the Antiplatelet Effects Comparing Ticagrelor (Ticag. - AZD6140) With Clopidogrel (Clop.) Responder and Non-responders
Acronym: RESPOND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5130C00030
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-08

CONDITIONS: Stable Coronary Artery Disease
Keywords: coronary artery disease (CAD); heart attack; stable angina
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Angina, Stable | interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aspirin + Ticagrelor
  Interventions: Drug: Ticagrelor; Drug: Aspirin
- 2 (Active Comparator): Aspirin + Clopidogrel
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor — Tablets, Oral, 90 mg; 180 mg loading dose followed by 90 mg twice daily for 2 weeks
  Arms: 1
Drug: Clopidogrel — (over encapsulated) capsule, Oral, 75 mg; 600 mg loading dose followed by 75 mg once daily for 2 weeks
  Other Names: Plavix
  Arms: 2
Drug: Aspirin — Tablets, Oral, 75 mg to 100 mg once daily. Aspirin obtained locally by the investigator, according to local practice. The dose remained constant throughout the study

SUMMARY:
The purpose of this study is to see how Ticagrelor, a new oral reversible anti-platelet medication, affects platelets. Anti-platelet agents are medications that block the formation of blood clots by preventing the clumping of platelets. Blood clots prevent us from bleeding, but when they form inside the arteries their formation is linked to a risk of medical problems such as heart attack and stroke. This study investigated the effect of Ticagrelor on inhibition of platelet aggregation compared with clopidogrel in patients previously identified as non-responsive to clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented stable Coronary Artery Disease (CAD) (stable angina, previous MI history, previous history of revascularization)
* Females of child bearing potential must have a negative pregnancy test prior to receiving study drug and be willing to use a hormonal contraceptive in addition to double barrier contraception

Exclusion Criteria:

* History of Acute Coronary Syndromes within 12 months of screening or need for revascularization (angioplasty or coronary artery bypass graft (CABG))
* Any acute or chronic unstable condition in the past 30 days
* Have increased bleeding risk, eg, recent gastrointestinal bleed, uncontrolled high blood pressure, low platelet count, recent major trauma
* History of intolerance or allergy to aspirin or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Horrow, MD, Study Director — AstraZeneca; Paul Gurbel, md, Principal Investigator — Platelet & Thrombosis Research, LLC
Locations (10):
- United States (4):
  - Research Site, Jonesboro, Arkansas
  - Research Site, Ormond Beach, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Cincinnati, Ohio
- Canada (2):
  - Research Site, Hamilton, Ontario
  - Research Site, Lachine
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Esbjerg
- Research Site, Sheffield, United Kingdom

REFERENCES:
- [Derived] Jeong YH, Bliden KP, Antonino MJ, Park KS, Tantry US, Gurbel PA. Usefulness of the VerifyNow P2Y12 assay to evaluate the antiplatelet effects of ticagrelor and clopidogrel therapies. Am Heart J. 2012 Jul;164(1):35-42. doi: 10.1016/j.ahj.2012.03.022. Epub 2012 Jun 13. PMID 22795280
- [Derived] Jeong YH, Bliden KP, Tantry US, Gurbel PA. High on-treatment platelet reactivity assessed by various platelet function tests: is the consensus-defined cut-off of VASP-P platelet reactivity index too low? J Thromb Haemost. 2012 Mar;10(3):487-9. doi: 10.1111/j.1538-7836.2011.04604.x. No abstract available. PMID 22212857
- [Derived] Tantry US, Bliden KP, Wei C, Storey RF, Armstrong M, Butler K, Gurbel PA. First analysis of the relation between CYP2C19 genotype and pharmacodynamics in patients treated with ticagrelor versus clopidogrel: the ONSET/OFFSET and RESPOND genotype studies. Circ Cardiovasc Genet. 2010 Dec;3(6):556-66. doi: 10.1161/CIRCGENETICS.110.958561. Epub 2010 Nov 15. PMID 21079055
- [Derived] Gurbel PA, Bliden KP, Butler K, Antonino MJ, Wei C, Teng R, Rasmussen L, Storey RF, Nielsen T, Eikelboom JW, Sabe-Affaki G, Husted S, Kereiakes DJ, Henderson D, Patel DV, Tantry US. Response to ticagrelor in clopidogrel nonresponders and responders and effect of switching therapies: the RESPOND study. Circulation. 2010 Mar 16;121(10):1188-99. doi: 10.1161/CIRCULATIONAHA.109.919456. Epub 2010 Mar 1. PMID 20194878

RESULTS

PARTICIPANT FLOW:
Groups:
- Clopidogrel Non-responders - Clopidogrel to Ticagrelor: Non-responder definition: patients with an absolute difference of less than or equal to 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist. Clopidogrel 600 mg loading dose followed by 75 mg once daily (od) for 2 weeks; switch to ticagrelor 180 mg loading dose followed by 90 mg twice daily (bd) for 2 weeks.
- Clopidogrel Non-responders - Ticagrelor to Clopidogrel: Non-responder definition: patients with an absolute difference of less than or equal to 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist. Ticagrelor 180 mg loading dose followed by 90 mg twice daily (bd) for 2 weeks; switch to clopidogrel 600 mg loading dose followed by 75 mg once daily (od) for 2 weeks.
- Clopidogrel Responders - Clopidogrel to Clopidogrel: Responder definition: patients with an absolute difference greater than 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist. Clopidogrel 600 mg loading dose followed by 75 mg once daily (od) for 2 weeks; stay on clopidogrel 75 mg once daily (od) for 2 weeks
- Clopidogrel Responders - Clopidogrel to Ticagrelor: Responder definition: patients with an absolute difference greater than 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist. Clopidogrel 600 mg loading dose followed by 75 mg once daily (od) for 2 weeks; switch to ticagrelor 180 mg loading dose followed by 90 mg twice daily (bd) for 2 weeks.
- Clopidogrel Responders - Ticagrelor to Clopidogrel: Responder definition: patients with an absolute difference greater than 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist. Ticagrelor 180 mg loading dose followed by 90 mg twice daily (bd) for 2 weeks; switch to clopidogrel 600 mg loading dose followed by 75 mg once daily (od) for 2 weeks.
- Clopidogrel Responders - Ticagrelor to Ticagrelor: Responder definition: patients with an absolute difference greater than 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist. Ticagrelor 180 mg loading dose followed by 90 mg twice daily (bd) for 2 weeks; stay on ticagrelor 90 mg twice daily (bd) for 2 weeks.
Period: Overall Study
Arm/Group | Clopidogrel Non-responders - Clopidogrel to Ticagrelor | Clopidogrel Non-responders - Ticagrelor to Clopidogrel | Clopidogrel Responders - Clopidogrel to Clopidogrel | Clopidogrel Responders - Clopidogrel to Ticagrelor | Clopidogrel Responders - Ticagrelor to Clopidogrel | Clopidogrel Responders - Ticagrelor to Ticagrelor
Started | 20 | 21 | 13 | 16 | 14 | 14
Completed | 17 | 17 | 13 | 15 | 13 | 13
Not Completed | 3 | 4 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 2 | 3 | 0 | 0 | 0 | 1
Not completed — Developement of discontinuation criteria | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Severe Non-compliance to protocol | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clopidogrel Non-responders - Clopidogrel to Ticagrelor; Clopidogrel Non-responders - Ticagrelor to Clopidogrel: Non-responder definition: patients with an absolute difference of less than or equal to 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist
- Clopidogrel Responders - Clopidogrel to Clopidogrel; Clopidogrel Responders - Clopidogrel to Ticagrelor; Clopidogrel Responders - Ticagrelor to Clopidogrel; Clopidogrel Responders - Ticagrelor to Ticagrelor: Responder definition: patients with an absolute difference greater than 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist
- Total: Total of all reporting groups
Arm/Group | Clopidogrel Non-responders - Clopidogrel to Ticagrelor | Clopidogrel Non-responders - Ticagrelor to Clopidogrel | Clopidogrel Responders - Clopidogrel to Clopidogrel | Clopidogrel Responders - Clopidogrel to Ticagrelor | Clopidogrel Responders - Ticagrelor to Clopidogrel | Clopidogrel Responders - Ticagrelor to Ticagrelor | Total
Number analyzed (Participants) | 20 | 21 | 13 | 16 | 14 | 14 | 98
Age Continuous [Mean (Standard Deviation); unit: year] | 67.25 (8.12) | 64.57 (6.31) | 65.46 (8.68) | 64.56 (8.56) | 63.21 (9.23) | 61.57 (8.22) | 64.8 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 3 | 2 | 3 | 1 | 22
  Male | 15 | 13 | 10 | 14 | 11 | 13 | 76

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Clopidogrel Non-responders Who Responded to Clopidogrel or Ticagrelor. - Comparing Ticag. (Day 28 of Clop. to Ticag., and Day 14 of Ticag. to Clop.) Versus Clop. (Day 14 of Clop. to Ticag., and Day 28 of Ticag. to Clop.)
Description: The primary definition of response to treatment is IPA >10% post treatment. The response is reported as percentage of participants of each treatment. Please refer to the protocol section for details about the interventions administered. IPA(%)=(PAb-PAt)/PAb*100. PA (platelet aggregation) is measured by LTA (Light Transmittance Aggregometry). PAb is the response at baseline (last measurement before study drug) and PAt is a response at post-treatment. IPA=0% means no PA inhibition and 100% means 100% PA inhibition.
Time Frame: Day 14 and Day 28, 4 Hrs Post Dose.
Population: Intent-to-treat analysis set: included patients who were assigned to a cohort, randomised to a treatment group, received at least one dose of study drug, and contributed post baseline data. 32 subjects had IPA data; but 1 subject missing a treatment arm, did not qualify for McNemar's test.
Measure: Number; unit: Percent of Participants
Groups:
- Non-responder: Ticagrelor; Non-responder: Clopidogrel: patients with an absolute difference of less than or equal to 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist
Arm/Group | Non-responder: Ticagrelor | Non-responder: Clopidogrel
Number analyzed (Participants) | 31 | 31
Percent of Participants | 100 | 93.8

2. Primary Outcome: Proportion of Clopidogrel Non-responders Who Responded to Clopidogrel or Ticagrelor. - Comparing Ticag. (Day 28 of Clop. to Ticag., and Day 14 of Ticag. to Clop.) Versus Clop. (Day 14 of Clop. to Ticag., and Day 28 of Ticag. to Clop.
Description: The secondary definition of response to treatment is IPA >50% post treatment. The response is reported as percentage of participants of each treatment. Please refer to the protocol section for details about the interventions administered. IPA(%)=(PAb-PAt)/PAb*100. PA (platelet aggregation) is measured by LTA (Light Transmittance Aggregometry). PAb is the response at baseline (last measurement before study drug) and PAt is a response at post-treatment. IPA=0% means no PA inhibition and 100% means 100% PA inhibition.
Time Frame: Day 14, and day 28, 4 hours post dose
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Non-responder: Ticagrelor | Non-responder: Clopidogrel
Number analyzed (Participants) | 31 | 31
Percent of participants | 81.3 | 25.0

3. Secondary Outcome: Clopidogrel Responders Final Extent IPA Post Switching Treatment - Comparing Ticagrelor to Ticagrelor Versus Ticagrelor to Clopidogrel on Day 15
Description: IPA(%)=(PAb-PAt)/PAb*100. PA (platelet aggregation) is measured by LTA (Light Transmittance Aggregometry). PAb is the response at baseline (last measurement before study drug) and PAt is a response at post-treatment. IPA=0% means no PA inhibition and 100% means 100% PA inhibition. Please refer to the protocol section for details about the interventions administered.
Time Frame: Day 15, 4 hrs post switching
Population: Intent-to-treat analysis set: included patients who were assigned to a cohort, randomised to a treatment group, received at least one dose of study drug, and contributed post baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Responder: Ticagrelor; Responder: Clopidogrel: patients with an absolute difference greater than 10% between baseline and post-treatment platelet aggregation (maximum extent) with 20 μM ADP used as the agonist
Arm/Group | Responder: Ticagrelor | Responder: Clopidogrel
Number analyzed (Participants) | 12 | 10
Percent | 66.7 [49.7 to 83.7] | 65.3 [46.5 to 84.2]

4. Secondary Outcome: Clopidogrel Responders Final Extent IPA Post Switching Treatment - Comparing Ticagrelor to Ticagrelor Versus Ticagrelor to Clopidogrel on Day 28
Description: as for outcome 3
Time Frame: 4 hrs post first dose on day 28
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Responder: Ticagrelor | Responder: Clopidogrel
Number analyzed (Participants) | 11 | 10
Percent | 91.0 [77.1 to 104.9] | 61.2 [46.4 to 76.0]

5. Secondary Outcome: Clopidogrel Responders Final Extent IPA Post Switching Treatment - Comparing Clopidogrel to Clopidogrel Versus Clopidogrel to Ticagrelor on Day 15
Description: as for outcome 3
Time Frame: Day 15, 4 hrs post switching
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Responder: Ticagrelor | Responder: Clopidogrel
Number analyzed (Participants) | 14 | 13
Percent | 95.0 [87.7 to 102.4] | 48.5 [40.8 to 56.2]

6. Secondary Outcome: Clopidogrel Responders Final Extent IPA Post Switching Treatment - Comparing Clopidogrel to Clopidogrel Versus Clopidogrel to Ticagrelor on Day 28
Description: as for outcome 3
Time Frame: 4 hrs post first dose on day 28
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Responder: Ticagrelor | Responder: Clopidogrel
Number analyzed (Participants) | 14 | 13
Percent | 77.4 [67.0 to 87.8] | 60.8 [49.9 to 71.7]

ADVERSE EVENTS:
Time Frame: Switching Period - first 24 hrs (Day 15), patients switched study medication (from clop. to ticag. or vice versa). Non-Switching Period - Day 1-14 and Day 16-28.
Description: Analysis included all randomized subjects.
Groups:
- Clopidogrel Non-Responders/Non-Switching Period: Ticagrelor: included non-responders exposed to ticagrelor on Day 1-14, Day 16-28.
- Clopidogrel Non-Responders/Non-Switching Period: Clopidogrel: included non-responders exposed to clopidogrel on Day 1-14, Day 16-28.
- Clop. Non-Responders/Switching Period:Ticagrelor-Clopidogrel: included non-responders exposed to ticagrelor switching to clopidogrel on Day 15.
- Clop. Non-Responders/Switching Period: Clopidogrel-Ticagrelor: included non-responders exposed to clopidogrel switching to ticagrelor on Day 15.
- Clop. Responders/Non-Switching Period: Ticagrelor: included responders exposed to ticagrelor on Day 1-14, Day 16-28.
- Clop. Responders/Non-Switching Period: Clopidogrel: included responders exposed to clopidogrel on Day 1-14, Day 16-28.
- Clop. Responders/Switching Period: Ticagrelor-Clopidogrel: included responders exposed to ticagrelor switching to clopidogrel on Day 15.
- Clop. Responders/Switching Period: Clopidogrel-Ticagrelor: included responders exposed to clopidogrel switching to ticagrelor on Day 15.
Arm/Group | Clopidogrel Non-Responders/Non-Switching Period: Ticagrelor | Clopidogrel Non-Responders/Non-Switching Period: Clopidogrel | Clop. Non-Responders/Switching Period:Ticagrelor-Clopidogrel | Clop. Non-Responders/Switching Period: Clopidogrel-Ticagrelor | Clop. Responders/Non-Switching Period: Ticagrelor | Clop. Responders/Non-Switching Period: Clopidogrel | Clop. Responders/Switching Period: Ticagrelor-Clopidogrel | Clop. Responders/Switching Period: Clopidogrel-Ticagrelor
Serious Adverse Events (participants affected / at risk) | 2/39 | 0/38 | 0/18 | 0/18 | 2/44 | 0/42 | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 13/39 | 13/39 | 1/18 | 4/18 | 19/44 | 14/42 | 2/13 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clopidogrel Non-Responders/Non-Switching Period: Ticagrelor (N=39) | Clopidogrel Non-Responders/Non-Switching Period: Clopidogrel (N=38) | Clop. Non-Responders/Switching Period:Ticagrelor-Clopidogrel (N=18) | Clop. Non-Responders/Switching Period: Clopidogrel-Ticagrelor (N=18) | Clop. Responders/Non-Switching Period: Ticagrelor (N=44) | Clop. Responders/Non-Switching Period: Clopidogrel (N=42) | Clop. Responders/Switching Period: Ticagrelor-Clopidogrel (N=13) | Clop. Responders/Switching Period: Clopidogrel-Ticagrelor (N=16)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Clopidogrel Non-Responders/Non-Switching Period: Ticagrelor (N=39) | Clopidogrel Non-Responders/Non-Switching Period: Clopidogrel (N=39) | Clop. Non-Responders/Switching Period:Ticagrelor-Clopidogrel (N=18) | Clop. Non-Responders/Switching Period: Clopidogrel-Ticagrelor (N=18) | Clop. Responders/Non-Switching Period: Ticagrelor (N=44) | Clop. Responders/Non-Switching Period: Clopidogrel (N=42) | Clop. Responders/Switching Period: Ticagrelor-Clopidogrel (N=13) | Clop. Responders/Switching Period: Clopidogrel-Ticagrelor (N=16)
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0/38 | 0 | 0 | 1 | 4 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1/38 | 0 | 0 | 0 | 4 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 1/38 | 0 | 0 | 1 | 2 | 0 | 0
FATIGUE (General disorders) | 0 | 1/38 | 0 | 0 | 1 | 2 | 1 | 0
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 0 | 0/38 | 0 | 1 | 2 | 2 | 0 | 0
CHEST DISCOMFORT (General disorders) | 0 | 0/38 | 1 | 0 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0/38 | 0 | 0 | 3 | 0 | 0 | 0
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 2/38 | 0 | 0 | 2 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0/38 | 0 | 0 | 0 | 1 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1/38 | 0 | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 3/38 | 0 | 2 | 1 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 2 | 1/38 | 0 | 0 | 0 | 1 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 2/38 | 0 | 0 | 1 | 0 | 0 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 1/38 | 0 | 1 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 3/38 | 1 | 2 | 6 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0/38 | 0 | 0 | 3 | 0 | 0 | 0
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 3 | 1/38 | 0 | 0 | 2 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AZ for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites.